CLINICAL TRIAL: NCT07246265
Title: Morphine Clearance and Glomerular Filtration in Sickle Cell Patients in Crisis in Intensive Care
Acronym: PHEDREA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DR230314; 2024-511985-34-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-29; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease; Glomerular Hyperfiltration; Sickle Cell Nephropathy; Vaso-Occlusive Crises; Acute Chest Syndrome
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Acute Chest Syndrome | interventions — Glomerular Filtration Rate; Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Determination of glomerular filtration rate by Iohexol (Experimental): Four morphine dosages, and a precise determination of the glomerular filtration rate by the measure of the elimination rate of iohexol will be carried out. The investigators will analyse in which patients and for which glomerular filtration rate there is morphine underdosage and simultaneously evaluate the effectiveness of analgesia and the amount of analgesics required.
  Interventions: Drug: Injection of iohexol for glomerular filtration rate (GFR) measurement

INTERVENTIONS:
Drug: Injection of iohexol for glomerular filtration rate (GFR) measurement — All patients will receive the same intervention. In included patients, 5 mL of iohexol will be injected, followed by blood sampling 5min, 1hr and 9hrs after iohexol injection for GFR measurement (as iohexol is known to be an exogenous maker for GFR measurement).
  Analgesia will be protocolized, based in particular on self-administered morphine (patient-controlled-analgesia). Morphine clearance will be measured thanks to 4 blood samples. Blood sampling for morphine and iohexol dosages will be synchronized in order to reduce the number of vascular punctures. Moreover, the first blood sample (5 minutes after iohexol injection) and the 4th blood sample for morphine dosage will be performed at the time of the daily biological analysis, still in order to reduce the number of vascular punctures. Thus, iohexol will be injected 5 minutes before the daily blood sampling for routine biological analysis.

SUMMARY:
Background: Sickle cell disease is a genetic disorder of haemoglobin (which carries oxygen in red blood cells). The shape of sickle cell-patients' red blood cells is abnormal. Thus, red blood cells can be blocked in small vessels, responsible for painful crises due to a lack of downstream circulation. These crisis (acute vaso-occlusive crisis) require strong treatment based on morphine, and often require intensive care.However, treatment is often insufficiently effective. Patient can also experiment acute chest syndrome, a complication of vaso-occlusive crisis, which can be responsible for respiratory failure. In addition, patients with sickle cell disease frequently have kidney damage called sickle cell nephropathy, which in the early stages of the disease is responsible for renal hyperfiltration, meaning that the kidneys filter the blood more than necessary, with faster elimination of drugs. For example, it is known that higher doses of antibiotics must be used in these patients than in the general population for the same effectiveness. The hypothesis of the study is that morphine, a drug eliminated by kidneys, is underdosed in patients with sickle cell disease, which is responsible for the difficulties in achieving sufficient analgesia.

Objective: To determine the glomerular filtration rate threshold for which it is necessary to prescribe higher doses of morphine in sickle cell patients with vaso-occlusive crisis.

Methods: inclusion of 100 patients admitted to intensive care for an acute vaso-occlusive crisis or acute chest syndrome and receiving morphine. Within 24 hours of study inclusion, four morphine dosages will be performed, in parallel with a precise determination of the glomerular filtration rate by measuring the elimination rate of a tracer, 100% eliminated by the kidneys and injected at the start of the study. This tracer is iohexol, a contrast agent commonly used in radiology. Morphine underdosage will be interpretated regarding glomerular filtration rate. The effectiveness of analgesia and the amount of analgesics required will be also be analyzed.

Outlook: At the end of this study, the investigators will be able to offer adapted doses of morphine for sickle cell patients in crisis, adapted to glomerular filtration rate, in the aim of personalizing analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Known homozygous sickle cell disease SS, SC, S-beta+, or S-beta0
* Admitted in an intensive care unit
* Clinical diagnosis of vaso-occlusive crisis and/or acute chest syndrome
* Receiving PCA treatment with morphine
* Patient's consent for study participation and/or from a relative if case of patient's incapacity
* Affiliation to social protection

Exclusion Criteria:

* Patient previously included in the study during a previous stay
* Injection of iodinated contrast medium outside the scope of the study within 24 hours prior to inclusion, or scheduled within 9 hours following the scheduled time of iohexol injection
* Contraindication to iohexol: known or suspected immediate or delayed hypersensitivity, thyrotoxicosis.
* Patient undergoing morphine treatment or substitution treatment such as methadone or buprenorphine prior to hospitalization (having received morphine or a derivative regardless of the route of administration in the week prior to hospitalization).
* Chronic liver disease likely to interfere with morphine metabolism (cirrhosis )
* Any condition that contraindicates the use of morphine according to the summary of product characteristics
* Patients under legal protection
* Pregnant or breastfeeding women

Exclusion criteria :

* Need for extrarenal epuration within 24 hours of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Therapeutic failure | 24 hours
  Prediction of therapeutic failure based on glomerular filtration rate according to the CKD-EPI formula (area under roc curve). Therapeutic failure is defined as a percentage of relief assessed by the verbal numerical scale not reaching 30% within 24 hours.
Glomerular filtration rate according to the CKD-EPI formula | 5 minutes
  Glomerular filtration rate according to the CKD-EPI formula

SECONDARY OUTCOMES:
Clearance of morphine and its metabolites M3G and M6G | 24 hours
  Correlation between clearance of morphine (and its metabolites M3G and M6G) and glomerular filtration rate according to the CKD-EPI formula.
Morphine dose administered | 24 hours
  Total dose of morphine administered during the day
Morphine dose administred | Day 7
  Total dose of morphine administered each day
Pain progression using the Visual Analog Scale | Every 4 hours for the first 7 days
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a 100-mm horizontal line ranging from 0 mm (no pain) to 100 mm (worst imaginable pain). Participants will indicate their pain level by marking a point on the line. Higher scores represent more severe pain. The change from baseline will be measured to assess pain progression.
Pain progression using a Numeric Rating Scale | Every 4 hours for the first 7 days
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (no pain) to 10 (worst imaginable pain). Participants verbally rate their pain on this numeric scale. Higher scores indicate worse pain.
Patient Global Impression of Change (PGIC) Over the First 7 Days | Daily, every 24 hours, from Day 1 to Day 7
  The Patient Global Impression of Change (PGIC) scale is a patient-reported outcome measure that assesses the patient's perception of change in their overall health status since the beginning of treatment. It is a 7-point Likert scale ranging from 1 (very much improved) to 7 (very much worse). Lower scores indicate a better outcome (improvement), while higher scores indicate worsening condition. PGIC will be assessed daily every 24 hours during the first 7 days of treatment.
Number of patients receiving paracetamol, nefopam, ketamine, NSAIDs, or nitrous oxide (MEOPA) within 24 hours | 24 hours
  The therapeutic regimen will be recorded by counting the number of patients who receive each of the following analgesics within the first 24 hours: paracetamol, nefopam, ketamine, non-steroidal anti-inflammatory drugs (NSAIDs), and nitrous oxide (MEOPA).
Adverse effects of morphine | Day 7
  Adverse effects of morphine include impaired alertness, bradypnea, hypercapnia, pruritus, constipation, bloating, nausea, vomiting, and acute urinary retention.
Glomerular filtration rate according to the CKD-EPI formula | 5 minutes
  Basal glomerular filtration rate according to the CKD-EPI formula and crisis glomerular filtration rate according to the CKD-EPI formula (5 minutes)
Plasma clearance of iohexol | 5 minutes, 1 hour et 9 hours
  Sample collection for iohexol dosage

OTHER OUTCOMES:
Age of participant at inclusion | Inclusion
  Age of the participant in years at the time of study inclusion. This variable will be analyzed to assess its correlation with therapeutic failure at 24 hours.
Socioeconomic Status According to EPICES (Evaluation de la précarité et des inégalités de santé dans les Centres d'examens de santé) Questionnaire | Inclusion
  Socioeconomic status will be assessed using the EPICES questionnaire, a validated tool to evaluate social deprivation. The score ranges from 0 (no deprivation) to 100 (maximum deprivation). This variable will be analyzed to assess its correlation with therapeutic failure at 24 hours.
Presence of chronic medical conditions at inclusion | Inclusion
  Documentation of chronic pathologies or comorbidities present at the time of inclusion, based on medical history and patient records. This variable will be analyzed to assess its correlation with therapeutic failure at 24 hours.
Number of vaso-occlusive crises or acute chest syndrome episodes requiring hospitalization in the previous year | Inclusion
  The number of hospitalizations due to vaso-occlusive crises or acute chest syndrome during the 12 months prior to inclusion. This variable will be analyzed to assess its correlation with therapeutic failure at 24 hours.
Number of unscheduled blood transfusions in the previous year | Inclusion
  The number of non-programmed blood transfusions received by the participant during the 12 months prior to inclusion. This variable will be analyzed to assess its correlation with therapeutic failure at 24 hours.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHRU de Tours, Tours, France
  - Henri-Mondor, Créteil
  - CH Le Mans, Le Mans
  - CHU de Nantes, Nantes
  - CHU d'Orléans, Orléans
  - CHU de Rennes, Rennes